CLINICAL TRIAL: NCT00381212
Title: A Pilot Study (Phase I/II) Testing the Immunologic Activity and Safety of AGS-004, an Autologous HIV Immunotherapeutic, in HIV-Infected Adults on HAART
Brief Title: A Pilot Study to Investigate the Safety and Immunologic Activity AGS-004 an Autologous HIV Immunotherapeutic Agent.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Université de Montréal (Other); Argos Therapeutics (Industry)
Responsible Party: Jean-Pierre Routy, MD, McGill University Health Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMB#06-003; CAN-HIV-001; CTN229
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: HIV Seropositivity; Acquired Immunodeficiency Syndrome
Keywords: Immunotherapeutic injection
MeSH Terms: conditions — HIV Seropositivity; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): AGS-004 immunotherapeutic injections.
  Interventions: Biological: AGS-004

INTERVENTIONS:
Biological: AGS-004 — Four intradermal injections of AGS-004-001 immunotherapeutic, 4 weeks apart.
  Other Names: AGS-004 immunotherapeutic

SUMMARY:
To Investigate the safety and immunologic activity of AGS-004, an autologous HIV Immunotherapeutic, in HIV-infected adults currently on stable antiretroviral therapy (ART) with durable viral suppression.

DETAILED DESCRIPTION:
Although an HIV infection can induce weak immune responses, current HIV immunotherapy using consensus antigens has not shown consistent clinical activity. The absence of clinical activity is associated with an inability to raise cytotoxic T lymphocytes (CTL) against HIV antigens and a failure to induce T cell memory. While strong immune responses may be generated to a consensus antigen, those responses do not offer antiviral protection against a patient's individual viral burden. The infecting virus' antigen variability likely prevents the establishment of effective CD4+ T cell memory and a strong CD8+ T cell effector arm.

We are investigating the induction of CTL responses in HIV-infected subjects by a novel HIV immunotherapeutic agent (AGS-004) in an effort to overcome the lack of polyvalent specificity of the immune response for autologous HIV antigens which has been one of the primary reasons for the failure of HIV immunotherapy to date.

This pilot study will investigate the safety and immunologic activity of AGS-004 an autologous HIV immunotherapeutic agent.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18 years and over,
* Documented HIV-1 infection,
* Durable viral suppression (≤ 200 copies HIV-1 RNA / mL) on first ART regimen for at least 12 weeks prior to entry,
* Availability of ≥ 2.5mL of continually-frozen plasma before starting ART (≥30,000 copies/mL),
* CD4+ T cell count ≥200 cells/mm3 at time of pre-ART sample,
* CD4+ T cell count of ≥350 cells/mm3 obtained within 4 weeks of study entry,

Exclusion Criteria:

* No co-infection with HBV or HCV,
* No history of lymph node irradiation or dissection,
* No prior use of any HIV vaccine,
* No use of hydroxyurea,
* No use of systemic corticosteroids or other non-permitted medications,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Immunologic activity of AGS-004 will be as measured by flow cytometry | 18 weeks

SECONDARY OUTCOMES:
To determine the safety of AGS-004 in the entire study population by frequency and severity of treatment emergent adverse events | 66 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Routy, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Immunodeficiency Service/Montreal Chest Institute, Montreal, Quebec, Canada